CLINICAL TRIAL: NCT02770079
Title: Botnia Clamp in Women Before, Immediately After Delivery and 6 Months Post Partum.
Brief Title: Insulin Sensitivity and Secretion During Pregnancy and Post Partum in Women With Gestational Diabetes.
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: GDM_Clamp_Skajaa
Record Dates: First submitted 2016-05-01; First posted 2016-05-12 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Diabetes, Gestational
Keywords: Insulin sensitivity
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood approximately 10 mL.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gestational diabetes: 10 women with gestational diabetes

SUMMARY:
Aim of the study:

To define insulin requirement during pregnancy and to identify the rapid changes in insulin sensitivity around parturition and the first 6 months post partum. Such knowledge would be clinically useful and markedly improve insulin treatment before and after parturition for women with type 1 diabetes and serve to identify the best possible timing of testing women with gestational diabetes mellitus (GDM) for the development of type 2 diabetes post partum.

Method:

Botnia clamp in women before, immediately after delivery and 6 months post partum. The investigators will compare 20 women with GDM in late pregnancy, day 15 post partum and 6 months post partum with 20 normal women investigated at the same time points. In addition the investigators will collect feces samples from the mother and baby in order to determine microbiota.

Perspectives:

Diabetes is a common condition with important implications for pregnancy outcome and long-term morbidity for mother and offspring. Accordingly, tailoring the best treatment is expected to have beneficial consequences both for the pregnant women and the future generation.

ELIGIBILITY:
Inclusion Criteria:

* Written consent before study start.
* Pregnant.
* GDM for the GDM group.
* No diabetes for the control group.

Exclusion Criteria:

* Women with multiple pregnancy.
* New pregnancy before all three examinations has been done.
* Severe, debilitating, concurrent diseases.
* Serious or intolerable adverse reactions associated with the studies.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All women visiting the outpatient gestational diabetes clinic at Aarhus University Hospital will be approached.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Determined one time between gestational week 32 to 37, 14 days postpartum and 6 months postpartum.
  Performing a Botnia clamp 3 times around parturition on women with GDM and comparing them with women with no GDM. The women will be their own control prospectively but also compared with a control group without gestational diabetes in order to compared them cross sectionally

SECONDARY OUTCOMES:
Changes in the microbiota | Determined one time between gestational week 32 to 37 (only the mother), 14 days postpartum and 6 months postpartum.
  Investigators will ask the participants to bring feces samples from themselves and their baby.

CONTACTS AND LOCATIONS:
Overall Officials: Per G Ovesen, MD, DMSc, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University Hospital, NBG, Aarhus, Denmark

REFERENCES:
- [Derived] Skajaa GO, Fuglsang J, Knorr S, Moller N, Ovesen P, Kampmann U. Changes in insulin sensitivity and insulin secretion during pregnancy and post partum in women with gestational diabetes. BMJ Open Diabetes Res Care. 2020 Oct;8(2):e001728. doi: 10.1136/bmjdrc-2020-001728. PMID 33115822